CLINICAL TRIAL: NCT00234247
Title: Study of the Long-term Outcomes of Nitric Oxide for Ventilated Premature Babies
Brief Title: Prolonged Outcomes After Nitric Oxide (PrONOx)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Derek C. Angus, MD, MPH, Chair, Critical Care Medicine, University of Pittsburgh
Other Study IDs: R01HL069991 (NIH); 1U01HL064857-01A1 (NIH)
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Lung Diseases; Bronchopulmonary Dysplasia; Premature Birth; Developmental Disabilities; Developmental Delay Disorders
MeSH Terms: conditions — Lung Diseases; Bronchopulmonary Dysplasia; Premature Birth; Developmental Disabilities

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Long Term Follow-Up — Extended and enhance the follow-up of the NHLBI iNO RCT by assessing the effects of iNO use on: 1.) long term clinical and childhood developmental outcomes; 2.) family impact, and; 3.) healthcare costs of prematurity-associated respiratory failure.

SUMMARY:
The purpose of this study is to look at the long term consequences of prematurity in infants treated with inhaled nitric oxide (iNO) while in the neonatal intensive care unit.

DETAILED DESCRIPTION:
Prematurity-associated respiratory failure is a growing public health problem. Although mortality has dropped with advances in perinatal care, this condition consumes considerable healthcare resources and is increasingly associated with worrisome long-term morbidity, developmental delay, and family burden. Inhaled nitric oxide (iNO), a selective pulmonary vasodilator that improves short-term outcomes in term neonates with respiratory failure, may benefit premature infants. Consequently, a NHLBI-funded randomized controlled trial (iNO RCT- NHLBI U01 HL064857) is assessing the effect of iNO on the combined end-point of mortality or oxygen dependency at 36 weeks post conceptional age in 800 infants with prematurity-associated respiratory failure.

However, prematurity-associated respiratory failure has a different etiology from respiratory failure in term infants and the wide array of long-term consequences that may be affected by iNO are not captured under the existing study design.

We therefore are extending and enhance the follow-up of the NHLBI iNO RCT. Specifically, we are assessing the effects of INO use on: #1. - long-term clinical and childhood developmental outcomes; #2. - family burden, and; #3. - healthcare costs of prematurity-associated respiratory failure. Under aim #4, we will use data from aims #1-3 to assess the cost-effectiveness of iNO in ventilated premature infants.

We are achieving these aims by augmenting the NHLBI iNO RCT data collection with: i.) survival follow-up for an average of 4 1/2 years; ii.) comprehensive, standardized follow-up clinic visits at 1, 2, 3 and 4 1/2 years to assess clinical outcomes, childhood development, and family burden; iii.) structured telephone interviews with parents every 3 months in year 1 and every 6 months thereafter for an average of 4½ years to assess chronic morbidity and post-discharge healthcare use; iv.) collection of detailed hospital bills for the primary hospitalization, and; v.) a comprehensive analysis plan.

This study will allow us to determine the long-term consequences of iNO therapy in this condition, aiding clinicians, families, and policymakers and immediately affecting care of critically ill infants. By combining with the NHLBI iNO RCT, we take advantage of an important opportunity to gather prospective long-term outcome data in a randomized fashion. Our proposal will significantly increase the return on investment in the RCT through a greater understanding of the impact of iNO therapy from a societal perspective. Neonatal intensive care has changed dramatically in the last ten years. This study will also provide contemporary information on the long-term outcomes of prematurity-associated respiratory failure following modern management. Finally, our data will allow assessment of the robustness of early proxies for subsequent outcomes, key for future study design in this area.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in "Inhaled NO for the Prevention of Chronic Lung Disease" trial (ClinicalTrials.gov Identifier: NCT00006401).

Exclusion Criteria:

* Did not consent to extended follow-up.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal intensive care patients - those with prematurity-associated respiratory failure following modern management.
Sampling Method: Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2002-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Assess the cost-effectiveness of iNO in ventilated premature infants using: long term clinical and childhood developmental outcomes; family impact; and healthcare costs of prematurity-associated respiratory failure | Five Years

CONTACTS AND LOCATIONS:
Overall Officials: Derek C Angus, MD, MPH, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CRISMA Laboratory Webpage- CRISMA coordinates the PrONOx study — http://www.ccm.upmc.edu/research/res_crisma.html